CLINICAL TRIAL: NCT05270278
Title: Characteristics of Type 2- High Inflammatory Endotype of Asthma Using New Biomarkers From Peripheral Blood and Exhaled Air and Its Effect on the Outcome of Therapy
Status: Completed | Type: Observational
Sponsor: Value Outcomes Ltd. (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: eNOSE; D3250L00044 (Other: AstraZeneca plc)
Record Dates: First submitted 2022-02-23; First posted 2022-03-08 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Asthma; Eosinophilic; Asthma Chronic; Bronchial Asthma; Asthma, Bronchial
Keywords: airway inflammation; airway obstruction; airway disease; serious asthma; pulmonary; biological therapy; omalizumab; dupilumab; mepolizumab; benralizumab; biomarkers; Exhaled Nitric Oxide Levels (FeNO); alveolar NO; cross-sectional study; exploratory analysis; conservative treatment
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma; Airway Obstruction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peripheral blood for evaluation of laboratory parameters
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1. Eosinophilic AB - initiated biological treatment against IL-5 or IL-5R: * initiated biological treatment - mepolizumab or benralizumab
  * judged by the treating physician, the patient cannot indicated treatment of type anti IgE or anti IL-4R
- 2. Eosinophilic AB - initiated biological treatment against IgE or IL-4R: * initiated biological treatment - omalizumab or dupilumab
  * judged by the treating physician, patient cannot indicated treatment type anti IL-5 or anti IL-5R
- 3. Eosinophilic AB - initiated biological treatment against IgE or IL-4R, or against IL-5 or IL-5R: * initiated biological treatment - omalizumab or dupilumab, or mepolizumab or benralizumab
  * judged by the treating physician, the patient could be potentially indicated to treatment with all 4 alternatives
- 4. Non-eosinophilic AB - without indication for biological treatment: * no biological treatment initiated
  * judged by the treating physician, the patient cannot be indicated to biological treatment

SUMMARY:
The goal of this study is to identify reliable, valid, easily measurable, interpretable, and useful biomarkers in peripheral blood and exhaled air by people with severe asthma for a more accurate description of the pathogenetic processes of asthma-related to the inflammatory endotype and the choice of biologic therapy.

DETAILED DESCRIPTION:
According to WHO, asthma bronchiale (AB) is the most frequent non-infectious disease in adults. There are 340 million patients with AB in the world. Approximately 500 000 patients in the Czech Republic are suffering from AB and 2,1 % have severe AB with the indication for conventional anti-inflammatory treatment. This subgroup of patients represents significantly high costs for the healthcare system.

There are many clinical phenotypes and molecular endotypes of AB and each of these groups has a different response to treatment. In the Czech republic is recommended classification into two main groups: eosinophil AB (type 2- high) and non-eosinophil AB (type 2- low). Eosinophil AB is furthered classified into two groups: eosinophil allergic (Th2-high) and eosinophil non-allergic (ILC2-high).

New biologicals, indicated for patients with the most severe form of AB, have entered the market during the last 15 years. These biologicals have confirmed their potential in randomized controlled studies. It can be assumed that there are 4 000 - 5000 patients suffering from this type of AB who could be indicated to this treatment in the Czech republic but, unfortunately, only 10 % of them have the access to such therapies in real practice.

Recommended markers of type 2- high AB don´t have strictly set critical values that are often unspecific, unstable in time, and often affected by other diseases or treatments. Some of the widely accepted predictors of response to biological treatment are eosinophilia, allergic reactivity, level of total and allergic-specific IgE, NO production in inhaled air (FeNO), gender, number of previous exacerbations, and duration of disease. Some of these predictors are used as decision criteria also in Global Initiative for Asthma (GINA) guidelines.

With respect to these facts, enormous efforts are being made worldwide to search for new biomarkers, which would be reliable, valid, easily measurable, interpretable, and useful for a more accurate description of the pathogenetic processes of asthma

ELIGIBILITY:
> Group 1 <

Inclusion Criteria:

* severe persistent eosinophilic AB (type 2- high)
* initiated biological treatment against IL-5 or IL-5R (mepolizumab, benralizumab) on this study visit
* judged by the treating physician, the patient cannot be indicated to treatment against anti IgE or anti IL-4R (omalizumab, dupilumab)
* signed informed consent
* signed consent to the processing of personal data
* willingness and ability to undergo examination

Exclusion Criteria:

* active smoker
* BMI higher than 40kg/m2
* ongoing oncological disease or oncological disease during the last 12 months
* severe cardiovascular disease
* uncontrolled diabetes mellitus
* contraindication of choosen biological treatment per SPC

  * Group 2 <

Inclusion Criteria:

* severe persistent eosinophil AB (type 2- high)
* initiated biological treatment against IgE or IL-4R (omalizumab, dupilumab) at this study visit
* judged by the treating physician, a patient cannot be indicated to treatment against anti IL-5 or anti IL-5R (mepolizumab, benralizumab)
* signed informed consent
* signed consent to the processing of personal data
* willingness and ability to undergo examination

Exclusion Criteria:

* active smoker
* BMI higher than 40kg/m2
* ongoing oncological disease or oncological disease during the last 12 months
* severe cardiovascular disease
* uncontrolled diabetes mellitus
* contraindication of choosen biological treatment per SPC

  * Group 3 <

Inclusion Criteria:

* severe persistent eosinophil AB (type 2- high)
* initiated biological treatment against IgE or IL-4R (omalizumab, dupilumab) or against IL-5 or IL-5R (mepolizumab, benralizumab) at this study visit was
* judged by the treating physician, the patient could be potentially indicated to treatment with all 4 alternatives
* signed informed consent
* signed consent to the processing of personal data
* willingness and ability to undergo examination

Exclusion Criteria:

* active smoker
* BMI higher than 40kg/m2
* ongoing oncological disease or oncological disease during the last 12 months
* severe cardiovascular disease
* uncontrolled diabetes mellitus
* contraindication of choosen biological treatment per SPC

  * Group 4 <

Inclusion Criteria:

* severe persistent non-eosinophil AB (type 2- low)
* judged by the treating physician, the patient cannot be indicated for biological treatment
* signed informed consent
* signed consent to the processing of personal data
* willingness and ability to undergo examination

Exclusion Criteria:

* active smoker
* BMI higher than 40kg/m2
* ongoing oncological disease or oncological disease during the last 12 months
* severe cardiovascular disease
* uncontrolled diabetes mellitus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients with severe AB type 2 - high (eosinophilic) and type 2- low (non-eosinophilic)
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Laboratory parameters (peripheral blood) - blood count | Baseline
Laboratory parameters (peripheral blood) - atopy | Baseline
Laboratory parameters (peripheral blood) - rheumatology | Baseline
  ANF, ENA, RF, ANCA (if not in the last 12 months)
Laboratory parameters (peripheral blood) - immunology | Baseline
  IgE, ECP, IgG, IgA, IgM, classes IgG
Laboratory parameters (peripheral blood) - flow cytometry (FACS) | Baseline
  The evaluation of eosinophil surface charakteristics per MFI
Clinical parameters (exhaled air) - FeNO | Baseline
Clinical parameters (exhaled air) - alveolar NO | Baseline
Clinical parameters (exhaled air) - eNOSE | Baseline
  The examination with "the electronical nose"

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Novosad, MUDr.,Ph.D., Principal Investigator — Fakultní nemocnice Hradec Králové
Locations (1):
- Fakultní nemocnice Hradec Králové, Hradec Králové, Královehradecký Kraj, Czechia